CLINICAL TRIAL: NCT04062422
Title: Prediction of Childhood Pulmonary Function Using Ulna Length in Children of Sub-saharian or Caribbean Ethnicity
Brief Title: Ulna Length in Black Children
Acronym: ULNOIR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: N°IDRCB 2017-A02962-51
Record Dates: First submitted 2019-08-19; First posted 2019-08-20 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2019-08

CONDITIONS: Ulna Length in Otherwise Healthy Children (With the Exception of Mild to Moderate Asthma)
Keywords: ulna; healthy children; height predicted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Height measurement is unreliable when neuromuscular weakness or spinal deformity is present. The aim of this study was to accurately predict pulmonary function from a limb segment (ulna) measurement that is precise and reproducible. Equations are available in caucasian children but are not available in children of sub-saharian or caribbean ethnicity, which was the aim of the study. To this end, 350 black children referred for pulmonary function testing for asthma follow-up will be included.

DETAILED DESCRIPTION:
Ulna (dominant and non-dominant arm), height measurement in 350 asthmatic children of sub-saharian or caribbean ethnicity (both parents). Repeatability analysis (ulna and height) for the first fifty children. Recording of pulmonary function tests results (spirometry, resistance measurements)

ELIGIBILITY:
Inclusion Criteria:

* age: 3 to 18 years old, two parents of sub-saharian or caribbean origin, referred for asthma suspicion or follow-up.

Exclusion Criteria:

* chronic disease excepting asthma, prematurity (<36 GW), steroid (>3/year), high dosage of inhaled steroid

Age Groups: Child, Adult, Older Adult
Study Population: child between 3 to 18 years old, two parents of sub-saharian or caribbean origin, referred for asthma suspicion or follow-up
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-04-28 (Actual)

PRIMARY OUTCOMES:
Ulna length | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Delclaux, PhD, Principal Investigator — APHP
Locations (1):
- Robert Debre Hospital, Paris, France

REFERENCES:
- [Result] Beydon N, Leye F, Bokov P, Delclaux C. Prediction of height using ulna length in African-Caribbean children. Pediatr Pulmonol. 2022 Sep;57(9):2032-2039. doi: 10.1002/ppul.25972. Epub 2022 May 21. PMID 35567383